CLINICAL TRIAL: NCT00670969
Title: Validation of Handheld Indirect Calorimeter in Overweight and Obese Patients
Brief Title: Validation of Hand Held Indirect Calorimeter in Overweight and Obese Patients
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 27265
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: People who will have the portable measurement taken first and handheld measurement taken second
- B: People who will have the handheld measurement taken first and portable measurement taken second

SUMMARY:
The purpose of this study is to determine, in a group of overweight or obese volunteers, if a handheld indirect calorimeter can accurately measures oxygen consumption to determine resting metabolic rate compared to a portable indirect calorimeter.

DETAILED DESCRIPTION:
1. Background and Rationale: With the growing number of overweight and obese Americans, health professionals need accurate and convenient tools to help personalize weight loss programs. Portable indirect calorimetry measurements are more expensive than handheld devices and often limited to research setting only, making them impractical for clinical use. Additionally equations used to estimate resting metabolic rate may be significantly inaccurate in overweight patients. Several studies have been conducted to determine the accuracy of handheld devices, however none have been done in the overweight and obese populations. If handheld calorimeters can accurately measure resting metabolic rate in overweight and obese patients, these tests may be used to improve and personalize weight management programs.
2. Key Objectives: To determine in a group of overweight or obese volunteers if a handheld indirect calorimeter can accurately measures oxygen consumption to determine resting metabolic rate.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years (no upper limit).
* Able to fast overnight.
* Have a BMI no less than 25 kg/m2.

Exclusion Criteria:

* All others

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Major Inclusion & Exclusion Criteria: Age at least 18 years (no upper limit). Able to fast overnight. Have a BMI no less than 25 kg/m2.
  Method of Identification of Subjects/Samples/Medical Records: Participants will be recruited with a flyer. Interested individuals will contact the investigators who will ask basic eligibility questions. If eligible, pre-test requirements will be explained to the participant (12 hour fast, avoidance of physical activity and smoking for the same time period.)
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2008-05; Primary Completion 2014-02-10 (Actual); Study Completion 2014-02-10 (Actual)

PRIMARY OUTCOMES:
Validate handheld calorimeter against a portable device | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Abigail E Schubert, MS, BA, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States